CLINICAL TRIAL: NCT07171918
Title: Prospective Observational Study to Determine the Utility of REMS in Comparison to NEWS2 for Predicting Morbidity and Mortality Among Patients Presenting to the ED Suspicion of Sepsis
Brief Title: Prospective Observational Study to Compare REMS vs NEWS2 for Patients Presenting to the ED With Sepsis
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr Reshma Haridas, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 38/22/IEC/JMMC&RI
Record Dates: First submitted 2023-07-14; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Anti-Bacterial Agents; Vasoconstrictor Agents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sepsis patients
  Interventions: Drug: Antibiotics, Vasopressors

INTERVENTIONS:
Drug: Antibiotics, Vasopressors — Both groups are scored on REMS and NEWS2, and then observed closely for the period of hospital stay with regard to ICU stay duration, ventilator days, vasopressor dependent days and total hospital duration

SUMMARY:
Prospective observational study to determine the utility of Rapid Emergency Medicine Score (REMS) in comparison to National Early Warning Score2 (NEWS2) for predicting morbidity and mortality among patients presenting to the Emergency Department with clinical suspicion of Sepsis

DETAILED DESCRIPTION:
Rapid Emergency Medicine Score (REMS) is an attenuated version of the Acute Physiology and Chronic Health Evaluation (APACHE) II score and has utility in predicting mortality in non- surgical patients. The NEWS2 can be used on all hospitalized patients to allow for the early detection of clinical deterioration and potential need for higher level of care. NEWS2 is closely associated with sepsis, however REMS is not so. But in recent studies comparing other EWS (Early Warning Scores) of sepsis, REMS was found to be superior.

Hence comparing REMs against NEWS2 to determine prognostication value of both scores in sepsis.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to ED of Tertiary Care Hospital in Thrissur.
* Patients age >/=18 years
* Patients who give informed consent for participation in the study.
* Suspicion of sepsis at the time of presentation to ED as per SSC Guidelines 2021

Exclusion Criteria:

* All patients with an alternate diagnosis other than sepsis at the time of discharge.
* Patients referred from other hospitals with diagnosis of sepsis, after initiation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the sensitivity of REMS score for predicting the morbidity and mortality as compared to NEWS2 in patients with clinical suspicion of sepsis as observed in earlier publications; citing hereby "The utility of the rapid emergency medicine score (REMS) compared with SIRS, qSOFA and NEWS for Predicting in-hospital Mortality among Patients with suspicion of Sepsis in an emergency department" & "NEWS2 Is Superior to qSOFA in Detecting Sepsis with Organ Dysfunction in the Emergency Department" with 95% confidence level & 15% relative allowable error, minimum sample size comes to 130.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the utility of REMS score over NEWS2 score - number of days of intensive care. | 18 months
  To compare REMS score against NEWS2 score with regard to morbidity indicators as - Number of days of intensive care
To determine the utility of REMS score over NEWS2 score - need for vasopressor administration | 18 months
  To compare REMS score against NEWS2 score with regard to morbidity indicators as - need for vasopressor administration
To determine the utility of REMS score over NEWS2 score - number of days spent as IP | 18 months
  To compare REMS score against NEWS2 score with regard to morbidity indicators as - number of days spent in hospital
To determine the utility of REMS score over NEWS2 score - need for mechanical ventilation | 18 months
  To compare REMS score against NEWS2 score with regard to morbidity indicators as - need for mechanical ventilation

SECONDARY OUTCOMES:
To determine in- hospital mortality of patients with clinical suspicion of sepsis | 30 days
  To compare the effectiveness of REMS and NEWS2 in predicting the in-hospital, 30 day mortality of patients admitted with clinical suspicion of sepsis.
To determine the utility of REMS score over NEWS2 score of patients admitted with qSOFA >/=2 | 18 months
  To compare the utility of REMS score over NEWS2 score for predicting the prognosis of patients admitted with qSOFA >/= 2 ; serum lactates >/= 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Jubilee Mission Medical College and Research Institute, Thrissur, India

IPD SHARING:
Plan to Share IPD: No